CLINICAL TRIAL: NCT02111460
Title: Multicentre Randomization Clinic Trial of Systemic Chemotherapy Combined With Loco-regional Radiotherapy vs. Chemotherapy Alone for Initially Untreated Distant Metastatic Nasopharyngeal Carcinoma With Chemosensitivity
Brief Title: Chemotherapy Combined With Radiotherapy vs Chemotherapy Alone for Distant Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC5010
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Initially; Untreated; Distant metastatic
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy (Experimental): Systemic Chemotherapy Combined with Loco-regional Radiotherapy
  Interventions: Radiation: Loco-regional Radiotherapy
- Chemotherapy (Active Comparator): Chemotherapy alone without Loco-regional Radiotherapy
  Interventions: Radiation: Loco-regional Radiotherapy

INTERVENTIONS:
Radiation: Loco-regional Radiotherapy — with or without Loco-regional Radiotherapy

SUMMARY:
This is a randomized parallel control trial to evaluate whether radical loco-regional Radiotherapy can prolong survival time of initial untreated metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The patients with initial untreated metastatic nasopharyngeal carcinoma
* Histologic diagnosis of nasopharyngeal carcinoma
* T1-4N0-3M1,IVC(according to the 7th AJCC edition)
* Aged between 18 and 65 years
* KPS≥70
* The therapeutic effect evaluation is CR or PR accomplished three course of cisplatin and 5-Fu
* Voluntary to participate and sign informed consent document

Exclusion Criteria:

* The patients suffered from serious neurologic disease
* Clinically significant cardiac, heart function less than or equal to 3 level
* Clinically significant respiratory disease,lung function less than or equal to 3 level
* Blood routine examination: WBC<3×109/L, Hemoglobin<90g/L, platelet count<75×109/L
* Abnormal liver function: total bilirubin or ALT or AST>2×ULN
* Abnormal renal function:serum creatinine>1.5×ULN
* Pregnant or lactating women
* The therapeutic effect evaluation is SD or PD accomplished three course of cisplatin and 5-Fu

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-10; Primary Completion 2019-08 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progress-free survival | 2 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site.
Complete Response (CR) | after the completion of the chemoradiotherapy treatment (up to 9 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the chemoradiotherapy treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only.

CONTACTS AND LOCATIONS:
Overall Officials: Ming y Chen, MD,Phd, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] You R, Liu YP, Huang PY, Zou X, Sun R, He YX, Wu YS, Shen GP, Zhang HD, Duan CY, Tan SH, Cao JY, Li JB, Xie YL, Zhang YN, Wang ZQ, Yang Q, Lin M, Jiang R, Zhang MX, Hua YJ, Tang LQ, Zhuang AH, Chen QY, Guo L, Mo HY, Chen Y, Mai HQ, Ling L, Liu Q, Chua MLK, Chen MY. Efficacy and Safety of Locoregional Radiotherapy With Chemotherapy vs Chemotherapy Alone in De Novo Metastatic Nasopharyngeal Carcinoma: A Multicenter Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1345-1352. doi: 10.1001/jamaoncol.2020.1808. PMID 32701129